CLINICAL TRIAL: NCT03305731
Title: Activating Behavior for Lasting Engagement After Stroke
Acronym: ABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Emily Kringle, Occupational Therapist, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO17070071
Record Dates: First submitted 2017-09-29; First posted 2017-10-10 (Actual); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Stroke; Physical Activity; Sedentary Lifestyle; Behavior, Health; Physical Disability
Keywords: Rehabilitation; Disability
MeSH Terms: conditions — Stroke; Motor Activity; Sedentary Behavior; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Activating Behavior for Lasting Engagement (Experimental): Participants will engage in the ABLE intervention.
  Interventions: Behavioral: Activating Behavior for Lasting Engagement

INTERVENTIONS:
Behavioral: Activating Behavior for Lasting Engagement — Activating Behavior for Lasting Engagement (ABLE) is a behavioral intervention in which participants learn skills to schedule, self-monitor, and problem solve strategies to overcome barriers to engagement in meaningful daily life activities.

SUMMARY:
Stroke survivors demonstrate high levels of sedentary behavior, placing them at risk for exacerbation of chronic health conditions. This may lead to recurrent stroke. Subtle cognitive impairments are common after stroke and can lead to difficulty self-monitoring and problem solving to overcome barriers to physical activity. Investigators developed the Activating Behavior for Lasting Engagement (ABLE) intervention to promote activity scheduling, self-monitoring, and problem solving activity over the full day. This study examines the effects of the ABLE intervention on sedentary behavior after stroke.

DETAILED DESCRIPTION:
The study advisory committee added a dose-matched, no-intervention delayed baseline to the study protocol following initial documentation of this study protocol on clinicaltrials.gov. The purpose of this delayed baseline design was to assess the baseline stability on the primary and secondary outcomes. The addition of this timepoint resulted in a shift of post-intervention timepoints as follows: Baseline 1 (week 1), Baseline 2 (week 6), Post-intervention (week 11), and Follow-up (week 18). Intervention was delivered between Baseline 2 and Post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of ischemic or hemorrhagic stroke
2. ≥6 months and ≤24 months post-stroke
3. ≥18 years of age
4. ambulatory in the community with or without an assistive device (e.g. walker, cane)
5. self-reported sedentary behavior (≥6 hours/day of sedentary behavior reported using the Sedentary Behavior Questionnaire)
6. reside within 50 miles of Pittsburgh, Pennsylvania

Exclusion Criteria:

1. severe aphasia (Boston Diagnostic Aphasia Examination score ≤1)
2. currently receiving outpatient or home care rehabilitation services (physical therapy, occupational therapy, or speech therapy)
3. current active cancer treatment
4. medical history of neurodegenerative disorder (i.e. dementia, Parkinson's disease, multiple sclerosis, Lou Gehrig's disease (ALS), glioblastoma, myasthenia gravis)
5. current major depressive disorder, psychiatric condition, substance abuse (Patient Health Questionnaire-9, PRIME-MD/MINI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily A Kringle, MOT, OTR/L, Principal Investigator — University of Pittsburgh; Elizabeth R Skidmore, PhD, OTR/L, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Activating Behavior for Lasting Engagement
Started (Baseline) | 21
Week 6 | 20
Week 11 | 20
Completed (Week 18) | 20
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Activating Behavior for Lasting Engagement
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.81 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Stroke Chronicity [Mean (Standard Deviation); unit: months] — Months elapsed between date of stroke onset and date of baseline testing. Date of stroke onset was extracted from medical records.
  months | 29.38 (14.34)
Stroke Type [Count of Participants; unit: Participants]
  Ischemic | 19
  Hemorrhagic | 2
Stroke Hemisphere [Count of Participants; unit: Participants]
  Left Hemisphere | 12
  Right Hemisphere | 7
  Both Hemispheres | 2
Prolonged Sitting [Mean (Standard Deviation); unit: minutes] — Measured using ActivPAL micro3 (Pal Technologies, Glasgow) following 7-day wear protocol. The mean daily duration of prolonged sitting accumulated in bouts of greater than or equal to 30 minutes was computed. Population: Non-compliance with activity monitor, n=1
  minutes
    number analyzed (Participants) | 20
    (all) | 466.56 (168.65)

OUTCOME MEASURES:

1. Primary Outcome: Change in Daily Sedentary Time Accumulated in Bouts Greater Than or Equal to 30 Minutes
Description: Objectively measured sedentary time (ActivPAL)
Time Frame: Baseline (Baseline=computed mean of week 1 and week 6) to 11 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Activating Behavior for Lasting Engagement
Number analyzed (Participants) | 20
minutes | 54.95 (81.10)

2. Primary Outcome: Change in Daily Number of Sedentary Breaks
Description: Objectively measured sedentary breaks (ActivPAL)
Time Frame: Baseline (Baseline=computed mean of week 1 and week 6) to 11 weeks
Measure: Mean (Standard Deviation); unit: breaks
Arm/Group | Activating Behavior for Lasting Engagement
Number analyzed (Participants) | 20
breaks | 2.61 (4.59)

3. Secondary Outcome: Change in Daily Number of Sedentary Breaks
Description: Objectively measured sedentary breaks (ActivPAL)
Time Frame: Baseline (Baseline=computed mean of week 1 and week 6) to 18 weeks
Measure: Mean (Standard Deviation); unit: breaks
Arm/Group | Activating Behavior for Lasting Engagement
Number analyzed (Participants) | 20
breaks | -2.55 (5.90)

4. Secondary Outcome: Change in Daily Sedentary Time Accumulated in Bouts Greater Than or Equal to 30 Minutes
Description: Objectively measured sedentary time (ActivPAL)
Time Frame: Baseline (Baseline=computed mean of week 1 and week 6) to 18 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Activating Behavior for Lasting Engagement
Number analyzed (Participants) | 20
minutes | 14.08 (58.95)

5. Secondary Outcome: Change in Participation
Description: Client rated participation in meaningful daily life activities using the Stroke Impact Scale - Participation Subscale
  The Stroke Impact Scale - Participation Subscale is a questionnaire-based measure of community participation. Participants rate their participation in 10 types of activities on a 1 to 5 point Likert-type scale. Scores are converted to a 0 to 100 scale, where low scores indicate low participation.
Time Frame: Baseline (Baseline=computed mean of week 1 and week 6) to 11 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activating Behavior for Lasting Engagement
Number analyzed (Participants) | 20
score on a scale | 1.48 (8.52)

6. Secondary Outcome: Change in Participation
Description: as for outcome 5
Time Frame: Baseline (Baseline=computed mean of week 1 and week 6) to 18 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activating Behavior for Lasting Engagement
Number analyzed (Participants) | 20
score on a scale | 1.33 (15.38)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Activating Behavior for Lasting Engagement
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT03305731/Prot_SAP_ICF_000.pdf